CLINICAL TRIAL: NCT01345786
Title: A 2-part, Cross-over Trial of NOMAC-E2 to Assess Bioequivalence Between the Phase 3 Pivotal Clinical Batches and a Batch Prepared Using the Commercial Drug Manufacturing Process
Brief Title: Bioequivalence of Nomegestrol Acetate (NOMAC) and Estradiol (E2) in Commercial Versus Phase 3 Pivotal Clinical Batches of NOMAC-E2 Tablets (P06328)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P06328
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy Postmenopausal Females

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Commercial NOMAC-E2, Part 1 (Experimental): Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2), either on the first day of Period 1 and Period 3 (for participants randomized to Sequence 1) or on the first day of Period 2 and Period 4 (for participants randomized to Sequence 2). Participants in Part 1 were from "Site 1".
  Interventions: Drug: Commercial NOMAC-E2
- Phase 3 NOMAC-E2, Part 1 (Active Comparator): Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch A"), either on the first day of Period 2 and Period 4 (for participants randomized to Sequence 1) or on the first day of Period 1 and Period 3 (for participants randomized to Sequence 2). Participants in Part 1 were from "Site 1".
  Interventions: Drug: Phase 3 NOMAC-E2 "Batch A"
- Commercial NOMAC-E2, Part 2 (Experimental): Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2), either on the first day of Period 1 and Period 3 (for participants randomized to Sequence 1) or on the first day of Period 2 and Period 4 (for participants randomized to Sequence 2). Participants in Part 2 were from "Site 2".
  Interventions: Drug: Commercial NOMAC-E2
- Phase 3 NOMAC-E2, Part 2 (Active Comparator): Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch B"), either on the first day of Period 2 and Period 4 (for participants randomized to Sequence 1) or on the first day of Period 1 and Period 3 (for participants randomized to Sequence 2). Participants in Part 2 were from "Site 2".
  Interventions: Drug: Phase 3 NOMAC-E2 "Batch B"

INTERVENTIONS:
Drug: Commercial NOMAC-E2 — 1 x 2.5 mg NOMAC/1.5 mg E2 fixed dose combination commercial tablet orally in the morning on Day 1 for all periods
  Other Names: SCH 900121
  Arms: Commercial NOMAC-E2, Part 1; Commercial NOMAC-E2, Part 2
Drug: Phase 3 NOMAC-E2 "Batch A" — 1 x 2.5 mg NOMAC/1.5 mg E2 fixed dose combination tablet from the Phase 3 clinical trial program ("Batch A") orally in the morning on Day 1 for all periods
  Other Names: SCH900121
  Arms: Phase 3 NOMAC-E2, Part 1
Drug: Phase 3 NOMAC-E2 "Batch B" — 1 x 2.5 mg NOMAC/1.5 mg E2 fixed dose combination tablet from the Phase 3 clinical trial program ("Batch B") orally in the morning on Day 1 for all periods
  Other Names: SCH 900121
  Arms: Phase 3 NOMAC-E2, Part 2

SUMMARY:
For the contraceptive application a film-coated tablet has been developed which combines nomegestrol acetate (NOMAC) with estradiol (E2). This was an open-label, randomized, single-dose, four-way, replicate, cross-over study design conducted in 2 parallel parts at two sites, one site per study part. The primary objective of Part 1 was to assess the bioequivalence of NOMAC and E2 of the drug product manufactured using the commercial process ("commercial batch") versus the Phase 3 drug product ("Batch A"). The primary objective of Part 2 was to assess bioequivalence of NOMAC and E2 of the drug product manufactured using the commercial process ("commercial batch") versus the Phase 3 drug product ("Batch B").

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy postmenopausal females between the ages of 45 and 70 years, inclusive, having a Body Mass Index (BMI) between 18 and 32, inclusive;
* Free of any clinically significant disease that would interfere with the study evaluations.

Key Exclusion Criteria:

* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug;
* History of any infectious disease that affected the subject's ability to participate in the trial;
* History of alcohol or drug abuse in the past 2 years;
* Previously received NOMAC-E2;
* Current participation in another clinical study or had participated in a clinical study (eg, laboratory or clinical evaluation) within 30 days of baseline;
* Smoked more than 10 cigarettes or equivalent tobacco use per day;
* History of malignancy;
* Contraindications for the use of contraceptive steroids;
* Recent history of medication use of certain medications specified in the protocol.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 - Sequence 1: Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2) on the first day of Period 1 and Period 3; Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch A") on the first day of Period 2 and Period 4. Participants in Part 1 were from "Site 1".
- Part 1 - Sequence 2: Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch A") on the first day of Period 1 and Period 3; Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2) on the first day of Period 2 and Period 4. Participants in Part 1 were from "Site 1".
- Part 2 - Sequence 1: Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2) on the first day of Period 1 and Period 3; Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch B") on the first day of Period 2 and Period 4. Participants in Part 2 were from "Site 2".
- Part 2 - Sequence 2: Participants received a single oral dose of the NOMAC-E2 fixed-dose combination tablet (2.5 mg NOMAC/1.5 mg E2) from the Phase 3 clinical trial program ("Batch B") on the first day of Period 1 and Period 3; Participants received a single oral dose of the NOMAC-E2 fixed-dose combination commercial tablet (2.5 mg NOMAC/1.5 mg E2) on the first day of Period 2 and Period 4. Participants in Part 2 were from "Site 2".
Period: Overall Study
Arm/Group | Part 1 - Sequence 1 | Part 1 - Sequence 2 | Part 2 - Sequence 1 | Part 2 - Sequence 2
Started | 41 (Number randomized) | 41 (Number randomized) | 38 (Number randomized) | 38 (Number randomized)
Treated | 41 | 41 | 37 | 37
Completed | 35 | 33 | 33 | 35
Not Completed | 6 | 8 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 3 | 1
Not completed — Subject withdrew consent | 2 | 2 | 1 | 0
Not completed — Noncompliance with protocol | 1 | 0 | 1 | 0
Not completed — Administrative | 3 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Sequence 1 | Part 1 - Sequence 2 | Part 2 - Sequence 1 | Part 2 - Sequence 2 | Total
Number analyzed (Participants) | 41 | 41 | 37 | 37 | 156
Age, Continuous [Mean (Full Range); unit: years] — Baseline characteristic is an overview of participants who received medication
  years | 55.3 [47 to 65] | 55.5 [45 to 70] | 55.9 [45 to 66] | 56.5 [46 to 70] | 55.78 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristic is an overview of participants who received medication
  Participants
    Female | 41 | 41 | 37 | 37 | 156
    Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration of NOMAC (Cmax of NOMAC)
Description: Bioequivalence for NOMAC and E2 were tested on the primary PK parameters: Cmax, AUC(infinity), and AUClast for NOMAC; and baseline adjusted AUC72 and Cmax for E2.
  Blood samples for pharmacokinetic (PK) evaluation of NOMAC were collected at predose (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 144 hours postdose Day 1.
Time Frame: 0 hours to time of maximum observed plasma concentration of NOMAC (tmax of NOMAC) (blood samples were collected for NOMAC evaluation up to 144 hours postdose)
Population: The # of plasma profiles analyzed is based on the # of single-dose administration periods actually completed (some participants discontinued without completing all 4 dosing periods).
  Part 1 analyses also excluded certain data from participants who were misdosed, and Part 2 analyses excluded participants who did not receive drug.
Measure: Mean (Full Range); unit: ng/mL
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
ng/mL | 6.22 [1.06 to 13.3] | 4.51 [1.72 to 11.6] | 8.03 [3.44 to 14.4] | 7.20 [2.70 to 12.6]
Statistical Analysis 1: Comparison: Commercial NOMAC-E2, Part 1 vs Phase 3 NOMAC-E2, Part 1; Test type: Non-Inferiority or Equivalence — Acceptance criteria of 80 - 125% were used for bioequivalence evaluations (bioequivalence concluded when 90% confidence interval fully contained within acceptance criteria); Ratio (Test/Ref %) = 137.5, 90% CI [131 to 144.4] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 2: Comparison: Commercial NOMAC-E2, Part 2 vs Phase 3 NOMAC-E2, Part 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 111.8, 90% CI [107.5 to 116.4] — Commercial Batch Test / Phase 3 Batch Reference

2. Primary Outcome: Baseline Corrected Maximum Observed Serum Concentration of E2 (Cmax of E2)
Description: Bioequivalence for NOMAC and E2 were tested on the primary PK parameters: Cmax, AUC(infinity), and AUClast for NOMAC; and baseline adjusted AUC72 and Cmax for E2.
  Blood samples for PK evaluation of E2 were collected predose (-1, -0.5, and 0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose Day 1; multiple predose samples were needed to correct for endogenous levels.
Time Frame: 0 hours to time of maximum observed serum concentration of E2 (tmax of E2) (blood samples were collected for E2 evaluation up to 96 hours postdose)
Population: as for outcome 1
Measure: Mean (Full Range); unit: pg/mL
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 138 | 137
pg/mL | 56.1 [10.2 to 1255] | 45.1 [9.76 to 324] | 44.4 [14.1 to 347] | 41.5 [19.8 to 133]
Statistical Analysis 1: Comparison: Commercial NOMAC-E2, Part 1 vs Phase 3 NOMAC-E2, Part 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 107.3, 90% CI [99 to 116.4] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 2: Comparison: Commercial NOMAC-E2, Part 2 vs Phase 3 NOMAC-E2, Part 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 103.6, 90% CI [99.2 to 108.2] — Commercial Batch Test / Phase 3 Batch Reference. In addition to the participants/profiles excluded, 1 participant from the Phase 3 Batch Reference group did not contribute to this comparison

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Measurable Sample (AUC Last) and Area Under the Concentration-time Curve From Time 0 to Infinity (AUC Infinity) for NOMAC
Description: Bioequivalence for NOMAC and E2 were tested on the primary PK parameters: Cmax, AUC(infinity), and AUClast for NOMAC; and baseline adjusted AUC72 and Cmax for E2.
  AUClast is the AUC from time 0 to the time of the final quantifiable sample.
  AUC infinity is the AUC from time 0 to infinity.
  Blood samples for PK evaluation of NOMAC were collected at predose (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 144 hours postdose Day 1.
Time Frame: 0 hours to time of the last measurable sample (blood samples were collected for NOMAC evaluation up to 144 hours postdose)
Population: as for outcome 1
Measure: Mean (Full Range); unit: ng*h/mL
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
ng*h/mL
  AUC last | 87.3 [9.71 to 151] | 78.1 [33.5 to 148] | 109 [45.4 to 207] | 106 [35.5 to 194]
  AUC infinity | 102 [13.6 to 182] | 93.3 [42.4 to 200] | 134 [49.2 to 299] | 131 [39.4 to 262]
Statistical Analysis 1: Comparison: Commercial NOMAC-E2, Part 1 vs Phase 3 NOMAC-E2, Part 1; Analysis for AUClast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 110.0, 90% CI [106.4 to 113.7] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 2: Comparison: Commercial NOMAC-E2, Part 2 vs Phase 3 NOMAC-E2, Part 2; Analysis for AUC last; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 103.3, 90% CI [100.9 to 105.7] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 3: Comparison: Commercial NOMAC-E2, Part 1 vs Phase 3 NOMAC-E2, Part 1; Analysis for AUC infinity; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 108.1, 90% CI [104.7 to 111.6] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 4: Comparison: Commercial NOMAC-E2, Part 2 vs Phase 3 NOMAC-E2, Part 2; Analysis for AUC infinity; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 103.1, 90% CI [100.5 to 105.8] — Commercial Batch Test / Phase 3 Batch Reference

4. Primary Outcome: Baseline Corrected Area Under the Concentration-time Curve From Time 0 to 72 Hours (AUC72) for E2
Description: Bioequivalence for NOMAC and E2 were tested on the primary PK parameters: Cmax, AUC(infinity), and AUClast for NOMAC; and baseline adjusted AUC72 and Cmax for E2.
  AUC72 is the AUC from time 0 to 72 hours.
  Blood samples for PK evaluation of E2 were collected predose (-1, -0.5, and 0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose Day 1; multiple predose samples were needed to correct for endogenous levels.
Time Frame: 0 hours to 72 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: pg*h/mL
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 137 | 138 | 137
pg*h/mL | 1315 [184 to 3132] | 1278 [140 to 3481] | 1359 [335 to 2813] | 1342 [297 to 3059]
Statistical Analysis 1: Comparison: Commercial NOMAC-E2, Part 1 vs Phase 3 NOMAC-E2, Part 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 101.5, 90% CI [96.7 to 106.4] — Commercial Batch Test / Phase 3 Batch Reference
Statistical Analysis 2: Comparison: Commercial NOMAC-E2, Part 2 vs Phase 3 NOMAC-E2, Part 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (Test/Ref %) = 101.3, 90% CI [98.1 to 104.7] — [estimate comment as in outcome 2, analysis 2]

5. Secondary Outcome: Tmax of NOMAC
Time Frame: 0 hours to tmax of NOMAC (blood samples were collected for NOMAC evaluation up to 144 hours postdose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
hours | 2 [0.5 to 6] | 2 [1 to 6] | 2 [1 to 6] | 2 [1 to 6]

6. Secondary Outcome: Tmax of E2
Time Frame: 0 hours to tmax of E2 (blood samples were collected for E2 evaluation up to 96 hours postdose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
hours | 6.02 [0.5 to 96] | 8 [0.5 to 96] | 8 [0.5 to 96] | 8 [0.5 to 24]

7. Secondary Outcome: Terminal Phase Half Life (t1/2) of NOMAC
Time Frame: 0 hours to t1/2 (blood samples were collected for NOMAC evaluation up to 144 hours postdose)
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
hours | 58.5 [17.3 to 137] | 61 [19.4 to 278] | 70.8 [23.5 to 201] | 69.9 [23.4 to 153]

8. Secondary Outcome: t1/2 of E2
Time Frame: 0 hours to t1/2 (blood samples were collected for E2 evaluation up to 96 hours postdose)
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 131 | 131 | 134 | 139
hours | 39.9 [8.3 to 855] | 39.1 [11.2 to 853] | 33.1 [9.02 to 94.8] | 34.6 [7.13 to 128]

9. Secondary Outcome: Clearance (Calculated for NOMAC Only)
Time Frame: blood samples were collected for NOMAC evaluation up to 144 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
L/h | 28.3 (16.1) | 29.9 (9.68) | 21.1 (7.96) | 22.1 (9.37)

10. Secondary Outcome: Volume of Distribution (Calculated for NOMAC Only)
Time Frame: blood samples were collected for NOMAC evaluation up to 144 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Units Other Than Participants: plasma profiles
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Number analyzed (Participants) | 70 | 71 | 72 | 72
Number analyzed (plasma profiles) | 138 | 138 | 140 | 140
L | 2208 (886) | 2445 (906) | 1988 (631) | 2061 (673)

ADVERSE EVENTS:
Description: Number of participants at risk for each group is the number of participants who received the treatment (batch).
Arm/Group | Commercial NOMAC-E2, Part 1 | Phase 3 NOMAC-E2, Part 1 | Commercial NOMAC-E2, Part 2 | Phase 3 NOMAC-E2, Part 2
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/77 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 44/80 | 35/77 | 36/72 | 35/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Commercial NOMAC-E2, Part 1 (N=80) | Phase 3 NOMAC-E2, Part 1 (N=77) | Commercial NOMAC-E2, Part 2 (N=72) | Phase 3 NOMAC-E2, Part 2 (N=72)
Constipation (Gastrointestinal disorders) | 5 (10) | 1 (2) | 8 (22) | 8 (20)
Nausea (Gastrointestinal disorders) | 5 (10) | 7 (14) | 3 (6) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (4) | 3 (6) | 6 (12)
Dizziness (Nervous system disorders) | 3 (8) | 5 (10) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 15 (40) | 14 (40) | 12 (26) | 13 (32)
Breast tenderness (Reproductive system and breast disorders) | 5 (10) | 3 (6) | 1 (2) | 2 (4)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 3 (6) | 8 (18)
Vaginal discharge (Reproductive system and breast disorders) | 4 (12) | 4 (10) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 5 (10) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (10) | 2 (4) | 4 (8)
Acne (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 8 (18) | 12 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 4 (8)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (8) | 1 (2)
Hot flush (Vascular disorders) | 14 (40) | 8 (20) | 9 (22) | 8 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide sponsor w/ review copies of abstracts or manuscripts for publication that report any results of the study, 45 days before submission for publication or presentation. The sponsor shall have the right to review/comment on the material. If the parties disagree about the appropriateness of the material, PI must meet with sponsor's representatives before submission for publication, for the purpose of making good faith efforts to discuss and resolve any issues of disagreement.